CLINICAL TRIAL: NCT04209296
Title: A Retrospective Chart Review of Patients Undergoing Ketamine Infusions at the Canadian Rapid Treatment Center of Excellence
Brief Title: Chart Review of Patients Undergoing Ketamine Infusions
Status: Completed | Type: Observational
Sponsor: Brain and Cognition Discovery Foundation (Other)
Responsible Party: Principal Investigator, Roger McIntyre, Chairman and Executive Director, Brain and Cognition Discovery Foundation
Other Study IDs: Pro00040593
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Obsessive-Compulsive Disorder; Post Traumatic Stress Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Major Depressive Disorder (MDD): DSM-5 Diagnosis of MDD
  Interventions: Drug: Ketamine Hydrochloride
- Bipolar Disorder: DSM-5 Diagnosis of Bipolar Disorder
  Interventions: Drug: Ketamine Hydrochloride
- Obsessive Compulsive Disorder (OCD): DSM-5 Diagnosis of OCD
  Interventions: Drug: Ketamine Hydrochloride
- Post-traumatic Stress Disorder (PTSD): DSM-5 Diagnosis of PTSD
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine, a N-methyl-D-aspartate (NMDA) receptor antagonist has been used for general anesthesia since the 1970s, however, reports and trials by the end of the twentieth century and onward using subanesthetic doses suggested robust and rapid antidepressant and anti-suicidal effects. Ketamine is available as a 50/50 racemic mixture of enantiomers (S)-ketamine and (R)-ketamine.

SUMMARY:
The Canadian Rapid Treatment Center of Excellence (CRTCE) is a healthcare facility principally focused on providing best practices of intravenous ketamine treatment to adult patients suffering from mental health conditions. The center focuses specifically on treating individuals suffering from major depression disorder, bipolar disorder, post-traumatic stress disorder and obsessive compulsive disorder as their primary diagnosis. Herein, this retrospective analysis aims to look at past data in order to further develop our understanding of ketamine in the use of psychiatry.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years old. Patients over the age of 65 must receive additional approval to ensure safety.
2. Diagnosed with either MDD, BD, PTSD or OCD by a healthcare provider.
3. Experiencing an MDE as defined and operationalized in the DSM 5.0.
4. Individuals who may have comorbid psychiatric conditions, but the comorbid psychiatric condition can be neither the primary condition or the primary clinical concern.
5. Individuals reporting suicidal ideation will be included, as suicidal ideation is a symptom of MDE.
6. Individuals must have received at least 2 guideline concordant treatment trials with pharmacotherapeutic treatment options as suggested in the CANMAT MDD guidelines 2016, Florida Medicaid guidelines 2017, or the CANMAT ISBD guidelines for BD 2013.
7. Individuals who have received ECT or other neuromodulatory treatments will be eligible for ketamine infusion.

Exclusion Criteria:

1. Individuals who meet DSM 5 criteria for a substance use and/or alcohol use disorder in the past 3 months.
2. Individuals who are experiencing psychotic symptoms as part of an MDE (mood congruent/mood incongruent).
3. Individuals who are unable to consent to the treatment.
4. Individuals who are unable to adhere to the protocol in its totality (i.e., remain in the clinic post infusion for up to 2-3 hours for observation).
5. Individuals who are unable to identify a person to assure their safe transport home following ketamine infusion.
6. Individuals with symptomatic traumatic brain injury.
7. Uncontrolled medical disorders (i.e., uncontrolled and/or insufficiently treated hypertension, allergies to ketamine and/or previous intolerability of ketamine).
8. Pregnancy.
9. Medical contraindications to ketamine.
10. Patients that are over 275 lbs

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators aim to analyze data from June 2018 (clinic opening) to present. Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Major Depressive Disorder (MDD), Bipolar Disorder (BD), Post-Traumatic Stress Disorder (PTSD) or Obsessive Compulsive Disorder (OCD) as determined by a psychiatrist. Patients must currently be experiencing a major depressive episode (MDE) as defined by the DSM-5.
Sampling Method: Non-Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology Self Report 16-Item | Over 4 inital infusions and maintance infusions (~2 years)
  The QIDS-SR16 is a self-report assessment used to evaluate depression severity in patients with a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, diagnosis of Major Depressive Episode. In total, there are 16 individual questions evaluating 9 DSM domains. The highest score is 27, indicating severe depression, while the lowest score is 0, which would suggest a complete absence of depressive symptoms.
Generalized Anxiety Disorder 7-item | Over 4 inital infusions and maintance infusions (~2 years)
  The GAD-7 is a 7 item self-report assessment used to evaluate symptoms of anxiety. The scale ranges from 0 (not at all) to 3 (nearly every day). To total score ranges from 0 suggesting a lack anxiety symptoms to 21, indicating severe anxiety.
Snaith-Hamilton Pleasure Scale | Over 4 inital infusions and maintance infusions (~2 years)
  The SHAPS assessment is a 14 item self report tool used to measure anhedonia. Each item can be have a response of 1 (Definitely agree), 2(Agree), 3(Disagree), and 4(definitely disagree). The total score ranges from 14 to 56, in which higher scores on the assessment indicate higher levels of anhedonia.
Sheehan Disability Scale | Over 4 inital infusions and maintance infusions (~2 years)
  The SDS contains 3 items, each ranging between zero to ten. The SDS is a self-reported assessment of disability within the context of depression. The total score ranges from 0, indicating no impairment, to 30, indicating severe impairment.
Endicott Work Productivity Scale | Over 4 inital infusions and maintance infusions (~2 years)
  The EWPS is a self report scale consisting of 25 items each ranging from 0 (high functioning) to 4 (low functioning). The total score ranges from 0 to 100, with 100 indicating extremely poor workplace productivity.

SECONDARY OUTCOMES:
Clinician Administered Dissociative States Scale | Over 4 inital infusions and maintance infusions (~2 years)
  The CADSS is a 23-item assessment administered by a clinician in order to evaluate dissociative symptoms. Each item is evaluated on a scale from 0, suggesting no dissociative symptom, to 4, suggesting extreme dissociation. In total, patients can score between 0 to 92, indicating extreme dissociation.

CONTACTS AND LOCATIONS:
Overall Officials: Roger S McIntyre, MD, Principal Investigator — Brain and Cognition Discovery Foundation
Locations (1):
- Canadian Rapid Treatment Centre of Excellence, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality. Only aggregate data will be published or made available.

REFERENCES:
- [Derived] Chisamore N, Danayan K, Rodrigues NB, Di Vincenzo JD, Meshkat S, Doyle Z, Mansur R, Phan L, Fancy F, Chau E, Tabassum A, Kratiuk K, Arekapudi A, McIntyre RS, Rosenblat JD. Real-world effectiveness of repeated intravenous ketamine infusions for treatment-resistant depression in transitional age youth. J Psychopharmacol. 2023 Aug;37(8):775-783. doi: 10.1177/02698811231171531. Epub 2023 May 16. PMID 37194253
- [Derived] Danayan K, Chisamore N, Rodrigues NB, Vincenzo JDD, Meshkat S, Doyle Z, Mansur R, Phan L, Fancy F, Chau E, Tabassum A, Kratiuk K, Arekapudi A, Teopiz KM, McIntyre RS, Rosenblat JD. Real world effectiveness of repeated ketamine infusions for treatment-resistant depression with comorbid borderline personality disorder. Psychiatry Res. 2023 May;323:115133. doi: 10.1016/j.psychres.2023.115133. Epub 2023 Mar 5. PMID 36889160
- [Derived] McIntyre RS, Rosenblat JD, Rodrigues NB, Lipsitz O, Chen-Li D, Lee JG, Nasri F, Subramaniapillai M, Kratiuk K, Wang A, Gill H, Mansur RB, Ho R, Lin K, Lee Y. The effect of intravenous ketamine on cognitive functions in adults with treatment-resistant major depressive or bipolar disorders: Results from the Canadian rapid treatment center of excellence (CRTCE). Psychiatry Res. 2021 Aug;302:113993. doi: 10.1016/j.psychres.2021.113993. Epub 2021 May 13. PMID 34034067
- [Derived] Lipsitz O, McIntyre RS, Rodrigues NB, Kaster TS, Cha DS, Brietzke E, Gill H, Nasri F, Lin K, Subramaniapillai M, Kratiuk K, Teopiz K, Lui LMW, Lee Y, Ho R, Shekotikhina M, Mansur RB, Rosenblat JD. Early symptomatic improvements as a predictor of response to repeated-dose intravenous ketamine: Results from the Canadian Rapid Treatment Center of Excellence. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Mar 8;105:110126. doi: 10.1016/j.pnpbp.2020.110126. Epub 2020 Oct 5. PMID 33031861